CLINICAL TRIAL: NCT06019572
Title: Long-term Outcomes After Surgery for Subaxial Cervical Spine Injuries in Octogenarians, a Matched Controlled Analysis
Brief Title: Spine Trauma in the Elderly
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Adrian Elmi Terander, Associate Professor, Karolinska Institutet
Other Study IDs: 4-1712/2021
Record Dates: First submitted 2023-08-25; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Spine Injury; Trauma; Surgery
MeSH Terms: conditions — Spinal Injuries; Wounds and Injuries | interventions — Laminectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Younger cohort (<80 years)
  Interventions: Procedure: Spine decompression and fixation surgery
- octogenarians (≥80 years)
  Interventions: Procedure: Spine decompression and fixation surgery

INTERVENTIONS:
Procedure: Spine decompression and fixation surgery — Surgery is performed by either an anterior or posterior approach. Anterior approach is performed with either discectomy or corpectomy accompanied fusion, while the posterior approach consist in a bilateral laminectomy accompanied by fusion.

SUMMARY:
Our study aims at investigating short and long-term outcomes following surgery for subaxial spine injuries in the elderly (octogenarian) population.

ELIGIBILITY:
Inclusion Criteria:

* All patients surgically treated for subaxial spine injuries between 2006 and 2018

Exclusion Criteria:

* Missing records

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study hospital is a publicly funded tertiary care center serving a region of approximately 2.3 million inhabitants and the region's only level 1 trauma center. Patients were identified through the surgical management software Orbit (Evry Healthcare Systems, Solna, Sweden).
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | 30-day postoperative period
  medical or surgical complications
Mortality | End of the study period (or end of data collection)
  death

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden